CLINICAL TRIAL: NCT00595855
Title: Deep Sclerectomy Versus Trabeculectomy. A 7 Year Prospective Randomised Clinical Trial
Brief Title: A Comparison Between Deep Sclerectomy and Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: STEFANO GANDOLFI, CHAIRMAN UNIV. EYE CLINIC, UNIVERSITY OF PARMA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARMASURG001
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Glaucoma
Keywords: glaucoma; surgery; non penetrating procedures; cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TE (Active Comparator): trabeculectomy
  Interventions: Procedure: trabeculectomy
- DS (Experimental): deep sclerectomy
  Interventions: Procedure: deep sclerectomy

INTERVENTIONS:
Procedure: trabeculectomy — Cairns-like trabeculectomy, limbus based, with 5_FU supplementation and argon laser suturelysis
  Arms: TE
Procedure: deep sclerectomy — deep sclerectomy with no implant and no sutures to the superficial flap, limbus based with suppplementation of FU (if needed)
  Arms: DS

SUMMARY:
Patients affected by medically uncontrolled open angle glaucoma will be randomised to either a non penetrating procedure (deep sclerectomy) or conventional trabeculectomy. The longterm efficacy (i.e. IOP w/out therapy) and safety (i.e. visual acuity, visual field stability and co-morbidities) will be evaluated.

DETAILED DESCRIPTION:
Prospective 7-year randomised investigator -masked clinical trial 79 eyes (79 patients) enrolled randomised to surgery by PEX and previous pilocarpine use Deep sclerectomy n = 41 Trabeculectomy n = 38 Estimated DS : TE success = 1:3 10% attrition ; power = 90%, alpha = 5%

Methods and evaluation of outcomes:

1. IOP: average of the two highest readings of the IOP phasing (6 readings)
2. VA: LogMAR (ETDRS chart)
3. Lens: LOCSII (slit lamp classification), worsening = one step progression confirmed at two visits

study visits: every 4 months

ELIGIBILITY:
Inclusion Criteria:

* Angle wide open
* Age > 65 yrs
* IOP > 23 and < 30 mmHg (average of the two highest readings of the daily IOP phasing)
* Topical beta blocker in fellow eye
* At least two medications in use + previous ALT
* MD < 20 dB (HFA 24-2 full threshold)
* LOCSII < C1-N1-P0

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 1997-10; Primary Completion 2007-01 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
intra ocular pressure without therapy (% of eyes within pre-selected cut-off limits) | 7 years

SECONDARY OUTCOMES:
(a) LogMAR visual acuity, (b) number of cataract extraction procedures | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Gandolfi Stefano, MD, Principal Investigator — University of Parma
Locations (1):
- Sally Williams, Parma, Italy